CLINICAL TRIAL: NCT04228016
Title: Efficacy of an Intranasal Stent on Nasal Obstruction at Night: A Prospective Multicenter Study
Brief Title: Efficacy of an Intranasal Stent on Nasal Obstruction at Night
Acronym: RHINASTENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Seven Dreamers Europe SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHINASTENT
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Device : nasal airway stent (Experimental): All patients consulting for predominantly nocturnal nasal obstruction who have benefited from Nasal Respiratory Functional Exploration with detection of pathological resistance in the decubitus.
  Interventions: Device: Device: nastent™

INTERVENTIONS:
Device: Device: nastent™ — Patients with Nasal obstruction at night, will be used intrasal stent during 15 nights. These are flexible silicone tubes that are lubricated and easy to insert into the nasal cavities, which would restore the permeability of the nasal cavities.

SUMMARY:
This study aims to demonstrate a decrease with normalization of nasal resistance in the forward decubital position and with an intra-nasal stent in patients with nasal obstruction.

DETAILED DESCRIPTION:
All patients consulting for nasal obstruction at night and who have functional nasal test with pathological resistance in decubitus position are included.

Functional nasal test (non invasive tests) will be performed before and after intranasal introduction of a stent: anterior rhinomanometry to measure nasal function by the measure of resistance and acoustic rhinometry to measure the geometry of nasal fossa by the measure of minimal sectional cross area sitting, after 30 minutes of decubitus then new measurements with a stent in decubitus position in each nostril .

ELIGIBILITY:
Inclusion Criteria:

1. Volontary patient
2. Over 18 years old or more.
3. Complain of a nasal obstruction more important (or only) at night (in decubitus position)

Exclusion Criteria:

1. Unability to sign the consent form
2. Allergy of stent component
3. Perforation of nasal septum
4. Haemostasis disorder or anticoagulant therapy
5. Bilateral obstructive septal deviation ou polyposis induce inability to introduce the stent in the nasal cavities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Nasal resistance in anterior rhinomanometry (sPa/ml/sec) | Day 15
  Change grom Baseline of Nasal resistance in anterior rhinomanometry. Sitting, lying in the meadow and Per stent nasal.

SECONDARY OUTCOMES:
Nasal Obstruction and Septoplasty Effectiveness (NOSE) | Day 15
  Scale [0-100] The higher the score, the more the quality of life is impaired.
Analog visual scale (EVA) of nocturnal nasal obstruction | Day 15
  Scale [0-10] The higher the score, the stronger the feeling of nasal obstruction.
Sino-Nasal Outcome Test 22 (SNOT-22) questionary | Day 15
  Scale [0-100]. The total score can range from 0 to 110, with values increasing as the severity of symptoms worsens
Epworth Sleepiness Scale (ESS) | Day 15
  Scale [0-24] The higher the score, the more the quality of life is impaired.
Compliance | Day 15
  Questionnaire on the use or non-use of the stent
Stent satisfaction | Day 15
  Number of patients satisfied with the stent
Stent tolerance | Day 15
  Questionnaire on stent tolerance or non-tolerance

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Intercommunal, Créteil, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No